CLINICAL TRIAL: NCT06788873
Title: Comparison of Elective Cervical Cerclage by Vaginal and by Laparoscopic Transabdominal Routes in the Periconceptional Period in the Patient with Unfavorable Obstetrical History
Brief Title: Comparison of Cervical Cerclage by Vaginal and by Laparoscopic Transabdominal Routes in the Periconceptional Period
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: ROUND-21
Record Dates: First submitted 2024-12-03; First posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-10

CONDITIONS: Cerclage, Cervical
Keywords: Vaginal cervical cerclage; Transabdominal cervical cerclage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Single pregnancy and vaginal cerclage: Participants with a single pregnancy and unfavorable obstetrical history (at least two preterm deliveries or abortions in the 2nd trimester of pregnancy) who underwent elective cervical cerclage vaginally between 01/01/2002 and 31/12/2020
  Interventions: Other: Data comparison
- No pregnancy and laparoscopic transabdominal cervical cerclage: Non-pregnant participants (with the same anamnestic characteristics as the first group) who underwent elective transabdominal laparoscopic cervical cerclage in the periconceptional period.
  Interventions: Other: Data comparison

INTERVENTIONS:
Other: Data comparison — For each participant, information will be collected on:
  * Gestational age at the time the cerclage was performed
  * Parity
  * Age
  * BMI
  * Ethnicity
  * Number of preterm deliveries
  * Gestational age of previous preterm deliveries
  * Previous uterine and/or cervix surgery (previous cerclage, conization, metroplasty, or other)
  * Type of cerclage performed
  * Operative times
  * Days of hospitalization
  * Surgical complications
  * Gestational age at the time of delivery
  * Mode of delivery (spontaneous, operative or cesarean)
  * Infant's weight at birth
  * Apgar at 1' and 5' minute
  * Ph newborn
  * Possible admission to neonatal intensive care unit.

SUMMARY:
The goal of this observational study is to compare two different surgical techniques of performing elective cervical cerclage in the prevention of preterm delivery, both of which are already widely used in common clinical practice: elective cervical cerclage by the vaginal route and laparoscopic transabdominal elective cervical cerclage.

DETAILED DESCRIPTION:
For the purpose of this study, no study-specific visits are planned. Data will be collected in a pseudo-anonymized manner, assigning each participant a sequence number.

For patients who undergo elective vaginal cervical cerclage at the division of Obstetrics and Prenatal Age Medicine or laparoscopic cerclage at the division of Gynecology and Human Reproductive Pathophysiology, the normal care pathway does not include additional follow-up visits for outpatient follow-up visits.

Regarding data collected in the past as part of the normal care pathway, patients will be asked to give informed consent in the context of a follow-up visit at which a practice staff member will be present.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unfavorable obstetric history, i.e., at least two previous preterm deliveries or second-trimester abortions who underwent elective prophylactic cervical cerclage (vaginal or laparoscopic) between 01/01/2002 and 31/12/2020
* Age ≥18 years
* Obtaining informed consent form
* Availability of clinical-demographic data

Exclusion Criteria:

* Multiple pregnancy

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants with single pregnancy (within 12- 14 weeks of amenorrhea) and unfavorable obstetrical history (at least two preterm deliveries or abortions in the second trimester of pregnancy) who between 01/01/2002 and 31/12/2020 who underwent elective cervical cerclage vaginally and non-pregnant patients (with the same anamnestic characteristics as the first group) who underwent elective transabdominal laparoscopic cervical cerclage in the periconceptional period.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of elective cervical cerclage vaginally and laparoscopic transabdominal elective cervical cerclage | up to 100 weeks
  The patients for whom such treatment is reserved are those with unfavorable obstetrical history (at least 2 preterm deliveries or abortions in the second trimester of pregnancy), who have an extremely high risk of recurrence.

SECONDARY OUTCOMES:
Comparison of maternal and fetal outcomes between the two groups | up to 100 weeks
  Live birth rate, gestational age at delivery, neonatal weight, and need for admission of the newborn to the Neonatal Intensive Care Unit (NICU).

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Montaguti, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy